CLINICAL TRIAL: NCT06186297
Title: Effect of a Cranberry Extract on Muscle Oxygenation and Mitochondrial Health in University Students
Brief Title: Boosting Performance: The Power of Cranberry Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Andreas Bergdahl, Associate Professor, Concordia University, Montreal
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 30017882
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Oxygen Consumption; Mitochondria; Blood Flow; Aerobic Capacity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry extract (Experimental)
  Interventions: Dietary Supplement: Cranberry extract
- Baseline (Active Comparator)
  Interventions: Dietary Supplement: Cranberry extract

INTERVENTIONS:
Dietary Supplement: Cranberry extract — polyphenol PAC-1

SUMMARY:
Cranberry is a fruit native to North America that is widely grown in Quebec and has been shown to have the highest antioxidant capacity among the most commonly eaten fruits. Consequently, consuming cranberries prior to exercising may help to improve exercise endurance by preventing accumulation of reactive oxygen species. For aerobic endurance, in order to maintain a certain pace for a long duration, runners need to effectively neutralize reactive oxygen species. Although it is not the only component involved in running, offsetting reactive oxygen species should improve running performance.

To test this, we plan to investigate the effects, both acute and chronic, of a cranberry extract on the oxygen consumption in 18-35 year old males and females.

The present research project will contribute to expand our knowledge of how cranberry extract can exert a positive effect, and thus improve aerobic performance or even every day life. This project can benefit a wide range of the population, from sedentary individuals and older adults to elite athletes by providing an all-natural supplement alternative.

DETAILED DESCRIPTION:
Each participant will be involved in the study for a period of 5 weeks, during which they will commit to 3 visits:

The first visit (on week 1) will be to obtain baseline measurements. During the second visit (on week 2), acute effects of the cranberry extract will be evaluated by giving a single high dose to the participants 1 hour before the trial events. The third visit (on week 5) will be to evaluate the chronic effects of the cranberry extract after 4 weeks of daily consumption. We will use the following instruments to gather data:

* Questionnaires (height, weight, dietary patterns, to determine training level, past injuries, single or multisport athlete etc.)
* Continuous wavelength NIRS will be used to measure oxygen levels in the quadriceps using portable Moxy monitors. For this test the subjects will be wearing the portable and convenient oxygen monitors taped firmly on the appropriate muscles. NIRS is a non-invasive method and measures the level of oxygenation in the muscle tissues by sending near-infrared light through the skin, which travels through the muscle fibers and is then recovered and returned to the surface of the skin and into the back of the sensor. As light moves through the skin layers (skin, fat and muscle), it scatters, and it identifies the oxygenated and the deoxygenated blood cells due to their colors. The blood cells identified are hemoglobin and myoglobin cells.

For the actual test, the quadriceps will be activated using electrical twitch stimulation at either 4 or 6Hz for 30 s at a current level that produce vigorous but submaximal contractions. During the contraction, the NIRS will be used in combination with short duration ischemic cuff periods (200 mmHg) applied by a Hokanson rapid cuff inflator. By repeating 5 second occlusion followed by 5 second deflation 6 times, at the same time as we activate the muscle, we will be able to determine muscle metabolism (mitochondrial oxygen consumption) by using the rate constant of the recovery from high to low metabolic rate.

• Skinfold measurement of the placement area for the Moxy oxygen monitors to determine if the light can penetrate subcutaneous tissues (has to be <15mm)

ELIGIBILITY:
Inclusion Criteria:

* recreationally active, healthy and between the ages of 18-35.

Exclusion Criteria:

* smoker; use of ergogenic substances or any kind or drugs that could alter the cardiovascular responses; resting BP higher than 140/90 mm Hg; and cardiovascular or metabolic disease (especially hypertension and diabetes)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | 20 minutes

SECONDARY OUTCOMES:
Blood flow | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No